CLINICAL TRIAL: NCT03082742
Title: The Effect of Thiazide and Loop Diuretic on Mineral and Bone Disorder in Chronic Kidney Disease Patients
Brief Title: The Effect of Diuretics on Mineral and Bone Disorder in Chronic Kidney Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Diuretics - CKD-MBD
Record Dates: First submitted 2017-02-27; First posted 2017-03-17 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: diuretics; furosemide; hydrochlorothiazide; CKD-MBD; HRpQCT; parathyroid hormone
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Hydrochlorothiazide; Furosemide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide (Active Comparator): Use of Furosemide, 40mg (1 tablet) per day, over 12 months
  Interventions: Drug: Furosemide
- Hydrochlorothiazide (Active Comparator): Use of Hydrochlorothiazide, 25mg (1 tablet) per day, over 12 months
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Hydrochlorothiazide
  Arms: Hydrochlorothiazide
Drug: Furosemide
  Arms: Furosemide

SUMMARY:
Chronic kidney disease (CKD) patients often have associated systemic hypertension due to volume retention, as one of the mechanisms, therefore the use of diuretics is widespread in this population. One of the major complications of CKD is mineral and bone metabolism disorder (CKD-MBD), which include changes in the levels of calcium, phosphorus, vitamin D deficiency, increased circulating levels of fibroblast growth factor (FGF-23) and parathyroid hormone (PTH). These alterations are responsible for fractures, cardiovascular disease and mortality among patients with CKD. According to diuretic mechanism of action, sometimes increasing serum calcium (in the case of furosemide), sometimes decreasing it (in the case of thiazide), it is expected that the serum calcium may be altered, even within the range of normality, with consequent impact on the levels of PTH. Although most studies have shown that the use of thiazide diuretics decreases the risk of fractures, some showed the opposite. Similarly, although most studies have shown increased risk of fracture in association to loop diuretics use, some have failed in demonstrated this outcome. Only one study, a cohort study in a population of CKD, showed that furosemide was directly related to increased calciuria and PTH levels and the use of thiazide, in turn, showed completely opposite effect. However, certain issues are still not completely solved, for example, the interference of renal function itself on calciuria. It is possible that calciuria is not a so simple explanation that justifies the PTH levels changes, as no correlation was seen between calciuria and PTH levels. Better understanding of the exact relationship between the use of diuretics and the impact on CKD-MBD may be an alternative intervention, easily accessible and relatively inexpensive. The purpose of this study is to evaluate the impact of diuretic, specifically hydrochlorothiazide and furosemide, on bone architecture and mineral metabolism.

DETAILED DESCRIPTION:
This is a prospective randomized study to test the effects of thiazide and furosemide in bone parameters, which will be assessed by peripheral micro-tomography at baseline and 12 months later. The role of calciuria in these possible changes will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Estimated Glomerular Filtration Rate (calculated by CKD-EPI) between 30 and 60 ml/min

Exclusion Criteria:

* Diabetes;
* chronic use of: steroid, bisphosphonates and calcium carbonate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Parathyroid hormone (PTH) level. | 12 months
  Bone metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Rosilene M Elias, M.D., Ph.D, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No